CLINICAL TRIAL: NCT05663060
Title: Evaluation Study of the Intestinal Microbiota and Quality of Life in Patients Suffering From Irritable Bowel Syndrome Treated With Bifidice
Brief Title: Evaluation Study of the Intestinal Microbiota and Quality of Life in Patients Suffering From IBS Treated With Bifidice
Acronym: Bifidice01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3291
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2022-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): Probiotic
  Interventions: Drug: Probiotic Formula

INTERVENTIONS:
Drug: Probiotic Formula — Probiotic Formula

SUMMARY:
Irritable bowel syndrome is the most common functional gastrointestinal disease and is characterized by high prevalence and chronic course.The pathology has a strong impact on the quality of life of affected patients and on health and social costs, these related to reduced productivity.The scarce efficacy and heavy side effects of traditional therapies lead these patients to often resort to alternative or complementary therapies. From the evaluation of the evidence of various probiotic preparations and food supplements, the investigators have used a commercial preparation characterized by the presence of bifidobacteria which have demonstrated some efficacy in thinking of improving the quality of life of these patients to evaluate quality of life, ability productivity and trend of some indices of disease severity in a small number of patients. These preliminary data could represent a starting point for more in-depth evaluations, also with placebo-controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Diagnosis of IBS according to Rome IV criteria
* Mild to moderate disease, as measured by FBDSI
* Absence of signs and symptoms that may suggest organic damage and, if indicated, negative instrumental investigations (colonoscopy and/or imaging)
* Prescription of Bifidice, according to normal clinical practice
* Informed consent expressed in written form

Exclusion Criteria:

* Patients undergoing surgical resection of the stomach, gallbladder, small or large intestine
* History of inflammatory bowel disease
* Severe SII, measured by FBDSI
* Active peptic ulcer
* History of ischemic colitis
* Active infectious enteritis
* Diagnosed with hypo- or hyperthyroidism
* Need for pharmacological treatments for IBS, antibiotics, antidepressants and laxatives
* Therapy in progress with drug or supplements included in the list of those not allowed (Paragraph N: to be established)
* Any disease that may affect gastrointestinal function and could interfere with appropriate assessment of abdominal pain or discomfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Modification of teh intestinal microbiota | 12 months
  Analysis of faecal samples (Next Generation Sequencing analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No